CLINICAL TRIAL: NCT06684860
Title: Comparative Diagnostic Performance of Rapid Urease Test Versus Molecular Testing for Diagnosis of Helicobacter Pylori
Brief Title: RUT vs. Molecular Testing for H. Pylori
Status: Recruiting | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Professor, Soonchunhyang University Hospital
Other Study IDs: SCH-HP-2024-12
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: H.Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RUT group: The rapid urease test (RUT) was performed for diagnosis of H. pylori infection.
- Molecular test group: DPO-PCR testing was performed for diagnosis of H. pylori infection.

SUMMARY:
The rapid urease test (RUT) is frequently performed for diagnosis of Helicobacter pylori infection in clinical practice. The RUT is a simple and inexpensive method that utilizes a commercial kit containing urea and a pH indicator such as phenol red. In the presence of H. pylori urease, urea is hydrolyzed to ammonia, which raises the pH of the medium, and changes the color of the kit from yellow to magenta or pink. The sensitivity and specificity of RUT were reported to range between 80-100% and 97-99%, respectively. When endoscopy is performed, RUT is known as the first-line method used for H. pylori diagnosis. However, RUT is an indirect test method, and has the disadvantage of causing false positivity due to other urease-producing bacteria.

To date, gold standards for H. pylori diagnosis are culture and histological examination Because H. pylori is a rather fastidious and slow-growing bacterium, antimicrobial susceptibility testing using culture methods is time-consuming (10-14 days) and requires specific expertise. Recently, dual priming oligonucleotide (DPO)-based multiplex polymerase chain reaction (PCR) was developed to diagnose H. pylori infection. Moreover, molecular testing can identify point mutations related to clarithromycin resistance. It can be performed in a standard thermocycler and takes only 4 h to complete. The concordance rate between conventional clarithromycin susceptibility testing and DPO-PCR was excellent up to 95%. However, there was no comparison study between RUT and molecular testing for H. pylori diagnosis.

DETAILED DESCRIPTION:
The investigators aim to compare the diagnostic accuracy of the RUT and molecular testing, and identify clinical factors associated with the discordant results between the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Gastroscopy can be performed
* H. pylori test and pathological analysis can be performed

Exclusion Criteria:

* Age < 20 or > 80 years
* Anemia (serum hemoglobin level < 10 g/dL)
* Severe systemic disease
* Advanced chronic liver disease
* Use of certain medications, including proton pump inhibitors, H2- receptor antagonists, or antibiotics
* History of H. pylori eradication
* Drug allergy to antibiotics
* History of gastric surgery
* Recent history of upper gastrointestinal bleeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: H. pylori-infected patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Current H. pylori infection status | 1 day
  RUT or molecular testing

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Digestive Disease Center, Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No